CLINICAL TRIAL: NCT03427645
Title: Development of a Tailored Life-Sustaining Treatment Decision Support Intervention for Stroke Surrogate Decision Makers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Darin Zahuranec, Associate Professor of Neurology, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00118298; 1R21NR016332-01A1 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stroke
Keywords: surrogate decision maker
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Surrogate Arm (No Intervention): Usual care control group will complete baseline and follow-up questionnaires with standard decision making techniques. This group will not be asked to use the decision making tool.
- Surrogate Decision Tool Arm (Experimental): This group will complete a baseline questionnaire, then use the tool and complete follow up questionnaires.
  Interventions: Behavioral: Decision tool

INTERVENTIONS:
Behavioral: Decision tool — A tailored web-based stroke decision support intervention. This web-based tool will be developed for use by the surrogate decision maker during the acute stroke hospitalization and will be designed to facilitate high quality patient-centered decisions and minimize adverse effects on the surrogate.
  Other Names: tailored decision support intervention
  Arms: Surrogate Decision Tool Arm

SUMMARY:
The trial is testing an investigator-developed decision support tool for surrogate decision makers for stroke patients that are unable to make medical decisions for themselves.

A historical usual care control group will be enrolled during tool development. The tool will then be tested in surrogates of hospitalized stroke patients.

DETAILED DESCRIPTION:
Decision support tools, specifically recommended in the 2010 Affordable Care Act, have been shown to improve the quality of decisions and reduce burden on the decision maker in multiple clinical settings, yet almost none have focused on life-sustaining treatments in acute critical illness such as stroke. This study proposes a comprehensive frame shift in how the health care team and surrogates collaborate on decisions regarding life-sustaining treatments for acute illness, by developing a tailored web-based stroke decision support intervention. This web-based tool will be developed for use by the surrogate decision maker during the acute stroke hospitalization and will be designed to facilitate high quality patient-centered decisions and minimize adverse effects on the surrogate.

The two project phases are: 1) Decision support intervention development; and 2) Pilot testing in surrogates of hospitalized stroke patients. A novel ordinal prognostic model will be developed and incorporated into the tool.

The project expects 25 surrogate-patient pairs in the control group, and 25 surrogate-patient pairs in the intervention group, which equals a total of 100 subjects.

ELIGIBILITY:
Surrogates:

Inclusion Criteria:

* Self-identify as the surrogate decision maker for eligible patient
* Able to read and communicate in English without an interpreter
* Limited to one surrogate per patient

Exclusion Criteria:

* No prior relationship with patient
* Dementia or other cognitive or health condition that would impair their ability to participate

Patients:

Inclusion Criteria:

* Ischemic stroke or spontaneous intracerebral hemorrhage
* Impaired decisional capacity (per treating team)
* Enrolled on or before full hospital day 5
* Minimum illness severity (either):

  * National Institutes of Health Stroke Scale ≥ 10
  * Glasgow coma scale ≤12

Exclusion Criteria:

* No surrogate available for study procedures
* Already on comfort measures only
* Physician refuses to allow approach for consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Acceptability of the decision tool intervention | Immediately post-intervention
  The proportion of cases where the surrogate completes use of the tool with high acceptability using the Acceptability E-Scale. The Acceptability E-Scale is a 6-item scale. A score of 1 indicates a negative evaluation and 5 indicates a positive evaluation. A score of 3 indicates a neutral evaluation. An individual will be considered to have high acceptability if the average response across the 6 items is 4 or higher)

SECONDARY OUTCOMES:
Accuracy of the surrogate's prognostic estimate for functional recovery | Within approximately 5 days of admission
  Calculated as the absolute value of the difference between the surrogate's estimate of the probability (0-100%) of return to functional independence by 90 days and the model based estimate of modified Rankin of 0-2. Range of this measure will be 0-100.
Decisional Self Efficacy scale | Within approximately 5 days of admission
  11-item scale (a score of 0 indicates not at all confident and a 4 indicates very confident) with ordered categorical responses, converted to a 0-100 scale based on the average of the responses to each item. A score of 0 means extremely low self-efficacy and a score of 100 means extremely high self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Darin Zahuranec, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Chen EP, Arslanian-Engoren C, Newhouse W, Egleston D, Sahgal S, Yande A, Fagerlin A, Zahuranec DB. Development and usability testing of Understanding Stroke, a tailored life-sustaining treatment decision support tool for stroke surrogate decision makers. BMC Palliat Care. 2020 Jul 20;19(1):110. doi: 10.1186/s12904-020-00617-x. PMID 32689982